CLINICAL TRIAL: NCT07068932
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-4506 Injection in Patients With Malignant Tumors
Brief Title: A Clinical Study of SHR-4506 Injection in Patients With Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4506-101
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Malignant Tumors of Adults

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4506 Group (Experimental)
  Interventions: Drug: SHR-4506 Injection

INTERVENTIONS:
Drug: SHR-4506 Injection — SHR-4506 injection.

SUMMARY:
The study is being conducted to evaluate the safety and tolerability of SHR-4506 Injection in patients with malignant tumors and to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, any gender.
2. ECOG performance status 0-1.
3. Histologically or cytologically confirmed malignant tumor patients who have failed standard therapy, or are intolerant to standard therapy, or have no standard treatment available.
4. Adequate organ function.
5. Voluntary participation in this clinical trial, with full understanding of study procedures and ability to provide written informed consent.
6. Expected survival ≥12 weeks.
7. Patients in the dose-expansion phase must have measurable lesions.
8. Agreement to use contraception from the time of signing the informed consent to at least 60 days after the last dose of the investigational drug.

Exclusion Criteria:

1. Prior treatment with the same class of investigational drug.
2. Confirmed or suspected central nervous system (CNS) tumor involvement.
3. Uncontrolled tumor-related pain.
4. Active autoimmune disease, history of immunodeficiency (including primary or secondary, e.g., HIV infection), or autoimmune disorders requiring systemic therapy.
5. Clinically significant cardiovascular disease history.
6. Known hypersensitivity to any component of the investigational drug.
7. Major surgery or significant trauma within 4 weeks prior to the first dose of the investigational drug; diagnostic or superficial surgery within 7 days before the first dose; or planned major surgery during the study period.
8. Adverse events from prior therapy have not recovered to ≤ CTCAE Grade 1.
9. Severe infection within 4 weeks before the first dose, or active infection within 2 weeks.
10. History of cerebrovascular accident within 6 months before the first dose of the investigational drug.
11. Patients with other active malignancies within 2 years prior to the first dose or concurrent malignancies.
12. Patients with any other condition judged by the investigator that makes the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicities (DLTs) | Up to 21 days.
Maximum Tolerated Dose (MTD) | Up to 21 days.
Incidence and severity of adverse events (AEs) | Up to 90 days after the last dose.
Incidence and severity of serious adverse events (SAEs) | Up to 90 days after the last dose.

SECONDARY OUTCOMES:
Objective response rate (ORR) assessed by the investigator | Up to 3 years.
Objective tumor response duration (DoR) | Up to 3 years.
Disease control rate (DCR) | Up to 3 years.
Progression free survival (PFS) | Up to 3 years.
Overall survival (OS) | Up to 3 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided